CLINICAL TRIAL: NCT05371093
Title: A Phase 3 Randomized, Open-Label, Multicenter Study Evaluating the Efficacy of Axicabtagene Ciloleucel Versus Standard of Care Therapy in Subjects With Relapsed/Refractory Follicular Lymphoma
Brief Title: Study of Axicabtagene Ciloleucel Versus Standard of Care Therapy in Participants With Relapsed/Refractory Follicular Lymphoma
Acronym: ZUMA-22
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KT-US-473-0133; 2021-003260-28 (EudraCT Number); 2024-511594-30 (Other: European Medicines Agency)
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Relapsed/Refractory Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — axicabtagene ciloleucel; Cyclophosphamide; fludarabine; Lenalidomide; Rituximab; Doxorubicin; Vincristine; Prednisone; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Axicabtagene Ciloleucel (Experimental): Participants will receive cyclophosphamide 500 mg/m^2/day intravenously (IV) and fludarabine 30 mg/m^2/day IV lymphodepleting chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-cluster of differentiation (CD)19 chimeric antigen receptor (CAR) transduced autologous T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells will be administered.
  Interventions: Biological: Axicabtagene Ciloleucel; Drug: Cyclophosphamide; Drug: Fludarabine
- Standard of Care Therapy (Active Comparator): Participants will receive the investigator's choice of one of the following therapies/dosing schedules:
  * Rituximab plus lenalidomide (R^2) for 12 cycles (28-day cycle)
    * Cycle 1: lenalidomide 20 mg/day on Day 1 through Day 21; rituximab 375 mg/m^2 on Day 1, Day 8, Day 15, and Day 22
    * Cycle 2 through Cycle 5: lenalidomide 20 mg/day on Day 1 through Day 21; Rituximab 375 mg/m2 on Day 1
    * Cycle 6 through Cycle 12: lenalidomide 20 mg/day on Day 1 through Day 21
  * Rituximab plus cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) for 6 cycles (21-day cycle)
    * rituximab 375 mg/m^2 on Day 1
    * cyclophosphamide 750 mg/m^2 on Day 1
    * doxorubicin 50 mg/m^2 on Day 1
    * vincristine 1.4 mg/m^2 (maximum 2 mg) on Day 1
    * prednisone 40 mg/m^2 on Day 1 through Day 5
  * Rituximab plus bendamustine (BR) for 6 cycles (28-day cycle)
    * rituximab 375 mg/m^2 on Day 1
    * bendamustine 90 mg/m^2 on Day 1 and Day 2
  Interventions: Drug: Cyclophosphamide; Drug: Lenalidomide; Drug: Rituximab; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Bendamustine

INTERVENTIONS:
Biological: Axicabtagene Ciloleucel — A single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells
  Other Names: Yescarta®; axi-cel
  Arms: Axicabtagene Ciloleucel
Drug: Cyclophosphamide — Administered intravenously
Drug: Fludarabine — Administered intravenously
  Arms: Axicabtagene Ciloleucel
Drug: Lenalidomide — Administered orally
  Arms: Standard of Care Therapy
Drug: Rituximab — Administered intravenously
  Arms: Standard of Care Therapy
Drug: Doxorubicin — Administered intravenously
  Arms: Standard of Care Therapy
Drug: Vincristine — Administered intravenously
  Arms: Standard of Care Therapy
Drug: Prednisone — Administered orally
  Arms: Standard of Care Therapy
Drug: Bendamustine — Administered intravenously
  Arms: Standard of Care Therapy

SUMMARY:
The goal of this clinical study is test how well the study drug, axicabtagene ciloleucel, works in participants with relapsed/refractory follicular lymphoma

DETAILED DESCRIPTION:
Five years after the last study participant is randomized, participants who have received axicabtagene ciloleucel will transition to a separate Long-term Follow-up study (study KT-US-982-5968) to complete the remainder of the 15-year follow-up assessments.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically-confirmed follicular lymphoma (FL) (Grade 1, 2, or 3a)
* Relapsed/refractory (R/r) disease after first-line chemoimmunotherapy and high-risk disease with relapse or progression within 24 months of the initial course of chemoimmunotherapy (ie, POD24), Or r/r disease after ≥ 2 prior systemic lines of therapy
* Clinical indication for treatment.
* At least 1 measurable lesion per the Lugano Classification {Cheson 2014}
* Adequate renal, hepatic, pulmonary, and cardiac function

Key Exclusion Criteria:

* Presence of large B cell lymphoma or transformed FL
* Small lymphocytic lymphoma
* Lymphoplasmacytic lymphoma
* Full-thickness involvement of the gastric wall by lymphoma
* FL Grade 3b
* Prior CD19-targeted therapy
* Prior CAR therapy or other genetically modified T-cell therapy
* Uncontrolled fungal, bacterial, viral, or other infection
* Active Infection with human immunodeficiency virus, hepatitis B virus or hepatitis C virus
* History or presence of a clincially significant central nervous system (CNS) disorder.
* History of autoimmune disease
* Known history or CNS lymphoma involvement
* Cardiac lymphoma involvement
* History of clinically significant cardiac disease 6 months before randomization
* Neuropathy greater than grade 2
* Females who are pregnant or breastfeeding
* Individuals of both genders who are not willing to practice birth control
* Presence of any indwelling line or drain (eg, percutaneous nephrostomy tube, indwelling Foley catheter, biliary drain, G/J-tube, pleural/peritoneal/pericardial catheter, or Ommaya reservoirs). Dedicated central venous access catheters such as Port-a-Cath or Hickman catheter are permitted.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) as Assessed by Blinded Central Assessment per Lugano Classification | Up to 5 years
  PFS is defined as the time from randomization to disease progression or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 5 years
  OS is defined as the time from randomization to death from any cause.
Complete Response (CR) Rate as Assessed by Blinded Central Assessment per Lugano Classification | Up to 5 years
  CR rate is defined as the proportion of participants with best overall response of CR during the study prior to any subsequent off-protocol anti-follicular lymphoma (FL) therapy.
Objective Response Rate (ORR) as Assessed by Blinded Central Assessment per Lugano Classification | Up to 5 years
  Objective response rate is defined as the proportion of participants with best overall response of either a complete response or a partial response during the study prior to any subsequent off-protocol anti-FL therapy.
Duration of Response (DOR) as Assessed by Blinded Central Assessment per Lugano Classification | Up to 5 years
  DOR is defined as the time from first objective response to disease progression or death from any cause.
Duration of CR as Assessed by Blinded Central Assessment per Lugano Classification | Up to 5 years
  Duration of CR is defined as the time from first CR to disease progression or death from any cause.
Event Free Survival (EFS) as Assessed by Blinded Central Assessment per Lugano Classification | Up to 5 years
  EFS is defined as the time from randomization to the earliest date of disease progression, the initiation of subsequent off-protocol anti-FL therapy, or death from any cause.
Time to Next Treatment (TTNT) | Up to 5 years
  TTNT is defined as the time from randomization to the start of subsequent off-protocol anti-lymphoma therapy or death from any cause.
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Randomization up to 5 years plus 30 days
Percentage of Participants Experiencing Clinically Significant Changes in Safety Laboratory Values | Randomization up to 5 years plus 30 days
Percentage of Participants with Replication-competent Retrovirus in Blood Over time | Up to 5 years
Change From Baseline in the Global Health Status Quality of Life Scale of the European Organisation for Research and Treatment of Cancer-Quality of Life Questionnaire-30 (EORTC QLQ-C30) | Baseline, up to 5 years
  The EORTC-QLQ-C30 is a multi-item questionnaire measuring the following content five (5) multi-item functional scales, three (3) multi-item symptom scales, one (1) global health status scale, and one (1) global health-related quality of life (HRQoL) each scale is measured from 0 to 100 after a linear transformation. Higher scores for functioning scales and for the Global Health Status or Global HRQoL scales indicate a higher level of functioning and a better HRQoL respectively, whereas higher scores in symptom scales represent a higher level of symptoms.
Change From Baseline in the Physical Functioning Domain of the EORTC QLQ-C30 | Baseline, up to 5 years
  The EORTC-QLQ-C30) is a multi-item questionnaire measuring the following content five (5) multi-item functional scales, three (3) multi-item symptom scales, one (1) global health status scale, and one (1) global health-related quality of life (HRQoL) each scale is measured from 0 to 100 after a linear transformation. Higher scores for functioning scales and for the Global Health Status or Global HRQoL scales indicate a higher level of functioning and a better HRQoL respectively, whereas higher scores in symptom scales represent a higher level of symptoms.
Change From Baseline in the Global Health Status Quality of Life Scale of the Low Grade Non-Hodgkin Lymphoma-20 (NHL-LG20) | Baseline, up to 5 years
  The NHL-LG20 is is a 20-item supplement questionnaire that was specifically developed to assess HRQoL in participants with low-grade non-Hodgkin lymphomas (such as follicular lymphoma). The NHL-LG20 includes multi-item scales of symptom burden, physical condition/fatigue, worries/fears on health and functioning, and emotional impact; and is administered in conjunction with the EORTC QLQ-C30. Each scale is measured from 0 to 100 after a linear transformation. Higher scores for functional scales and for the global health status or global HRQoL scales indicate a higher level of functioning and a better HRQoL, whereas higher scores in symptom scales represent a higher level of symptoms.
Change From Baseline in the Physical Functioning Domain of the NHL-LG20 | Baseline, up to 5 years
  The NHL-LG20 is is a 20-item supplement questionnaire that was specifically developed to assess HRQoL in participants with low-grade non-Hodgkin lymphomas (such as follicular lymphoma). The NHL-LG20 includes multi-item scales of symptom burden, physical condition/fatigue, worries/fears on health and functioning, and emotional impact; and is administered in conjunction with the EORTC QLQ-C30. Each scale is measured from 0 to 100 after a linear transformation. Higher scores for functional scales and for the global health status or global HRQoL scales indicate a higher level of functioning and a better HRQoL, whereas higher scores in symptom scales represent a higher level of symptoms.
Changes From Baseline in the European Quality of Life Five Dimensions Five Levels Scale (EQ-5D-5L) | Baseline, up to 5 years
  The EQ-5D-5L questionnaire is a generic measure of health status that provides a simple descriptive profile and a single index value. The EQ-5D-5L comprises 2 components: a questionnaire covering 5 dimensions and a tariff of values based upon direct valuations of health states using a visual analog scale (VAS). Rating gets recorded on a vertical VAS in which the endpoints are labeled best imaginable health state is 100 (on the top) and worst imaginable health state is 0 (on the bottom). Higher scores of EQ VAS indicate better health.
Changes From Baseline in the Visual Analog Scale (VAS) Scores | Baseline, up to 5 years
  The EQ-5D-5L VAS is a 20-cm VAS for recording self-rated current HRQoL state and is used to describe the participants health status on the day of the assessment. The EQ-5D-5L VAS score is recorded by each participant for his or her current HRQoL state and scored 0 ("the worst health you can imagine") to 100 ("the best health you can imagine"). Higher scores indicate better health.

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (52):
- United States (12):
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - Stanford Health Care, Stanford, California
  - Moffitt Cancer Center, Tampa, Florida
  - The University of Kansas Hospital, Westwood, Kansas
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Novant Health Cancer Institute Hematology - Charlotte, Charlotte, North Carolina
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - TriStar Centennial Medical Center - Cell Processing, Nashville, Tennessee
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- France (11):
  - Hopital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - Hôpital Claude Huriez-CHU de Lille, Lille
  - Institut Paoli-Calmettes, Marseille
  - Hopital Saint Eloi, Montpellier
  - Hopital Pitie-Salpetriere, Paris
  - CHU Bordeaux - Hospital Haut-Leveque - Centre Francois Magendie, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - Hopital Pontchaillou - CHU Rennes, Rennes
  - Centre Henri Becquerel, Rouen
- Germany (2):
  - Universitatsmedizin Gottingen, Göttingen
  - Universitatsklinikum Koln Klinik I fur Innere Medizin, Würzburg
- Italy (6):
  - ASST Papa Giovanni XXIII, Bergamo
  - Azienda Ospedallero-Universitaria di Bologna Policlinico Sant'Orsola-Malpighi, Bologna
  - Fondazione IRCCS - Istituto Nazionale Tumori, Milan
  - Ospedale San Raffaele, Milan
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Istituto Clinico Humanitas-IRCCS, Rozzano
- Japan (5):
  - Hyogo Medical University Hospital, Hyōgo
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Tohoku University Hospital, Miyagi
  - Okayama University Hospital, Okayama
  - Osaka University Hospital, Osaka
- Spain (8):
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Instituto Catalan de Oncologia - Hospital Duran i Reynolds (ICO L'Hospitalet), Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
- United Kingdom (8):
  - University Hospital Birmingham NHS Foundation Trust, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - University College London Hospitals NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - The University Hospital Southampton NHS Foundation Trust, Southampton
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KT-US-473-0133